CLINICAL TRIAL: NCT00044473
Title: An Open-Label Study of Levofloxacin to Evaluate Bacteriologic Outcome in the Treatment of Children Who Are at Risk for Acute Otitis Media That is Difficult to Treat
Brief Title: A Study of the Effectiness and Safety of Levofloxacin in Treating Children With a Rapid and Severe Onset of Infection and Inflammation of the Middle Ear That is Difficult to Treat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002389
Record Dates: First submitted 2002-08-29; First posted 2002-09-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Otitis Media
Keywords: Otitis Media; Ear Diaeases; Levofloxacin; Quinolones
MeSH Terms: conditions — Otitis Media | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of the study is to assess the rate of elimination of bacteria by levofloxacin in middle ear fluid of children with a rapid and severe onset of infection and inflammation of the middle ear who are at high risk for infections that are difficult to treat.

DETAILED DESCRIPTION:
Rapid and severe onset of middle ear infection is a common bacterial infection in children. These infections, particularly when they occur early in life and are recurrent, are associated with considerable disease and can lead to increasingly serious infections. This is a multicenter study to determine the effectiveness of levofloxacin in eliminating bacteria in the middle ear fluid of children between 6 months and 5 years of age with a rapid and severe onset of infection and inflammation of the middle ear (who are at high risk for infections that are difficult to treat). The study consists of a 1-day screening period when patients will be tested for eligibility for the study; a 4 to 6-day treatment, blood collection, possible collection of fluid from the middle ear, and assessment period; and a post-treatment period to assess the status of the middle ear infection. All patients will receive levofloxacin 2 times daily (up to a maximum daily dose of 500 mg) mixed with liquid and taken by mouth for 10 days. Safety evaluations will include laboratory tests, physical examinations, vital sign measurements, and recording of adverse events, including any report of joint pain or signs and symptoms of joint disease. Effectiveness will be assessed by the rate of elimination of the bacteria identified at the start of the study and by signs and symptoms, as well as microscopic evidence that the patient is cured of the middle ear infection. The study hypothesis is that levofloxacin will be effective in eliminating bacteria in the middle ear fluid of children with a rapid and severe onset of infection and inflammation of the middle ear and who are at high risk for infections that are difficult to treat. Levofloxacin 10 milligrams/kilogram (mg/kg) 2 times daily (up to a maximum daily dose of 500 mg) mixed with liquid and taken by mouth for 10 days

ELIGIBILITY:
Inclusion Criteria:

* Patients with signs and symptoms of rapid onset of severe infection of the middle ear defined as: either fluid draining from the middle ear (with a minimum of 2 of the following: decreased or absent eardrum mobility seen on physical examination
* yellow or white discoloration of the eardrum
* opaque eardrum) and (a minimum of 1 of the following: ear pain within 24 hours of the start of the study including the child's unexpected tugging or rubbing of the ear
* marked redness of the eardrum
* distinct fullness or bulging of the eardrum) or rapid onset of severe drainage of pus from the external ear lasting less than 48 hours and not due to inflammation of the external ear
* At risk for difficult-to-treat middle ear infection defined as having a minimum of 1 of the following: recurrent middle ear infection (defined as >=3 episodes, including the current episode, of rapid onset of rapid onset of severe middle ear infection during the 6 months before the study or >=4 episodes, including the current episode, of rapid onset of rapid onset of severe middle ear infection during the year before the study), persistent middle ear infection defined by signs and symptoms of rapid onset of severe middle ear infection on the third day after starting any antibiotic treatment (with the exception of amoxicillin/clavulanate that included >=90 milligrams/kilograms/day [mg/kg/day] of amoxicillin)
* Currently taking antibiotic medication to prevent middle ear infection (must be discontinued when beginning the study)
* Completed treatment with an antibiotic intended to treat middle ear infection within 30 days before the start of the study.

Exclusion Criteria:

* Patients with a history of a previous sensitivity or serious adverse reaction to the type of antibiotic used in this study
* Tubes in place in the affected ear to allow drainage of fluid from the middle ear
* Requirement of antibiotic therapy that affects the whole body, other than the study drug
* A serious bacterial infection in addition to middle ear infection that may interfere with assessment of the patient's response to study medication
* Diagnosis of bacterial meningitis
* Abnormal kidney function, as determined by blood test (serum creatinine)
* History or presence of joint disease or disease of the tissues surrounding joints, or any other signs or symptoms in muscles or bones that may make it difficult to evaluate any future complaints concerning muscles or bones
* Chronic use of corticosteroids

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2002-11; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Rate of elimination of the disease-producing bacteria identified at the start of the study; signs and symptoms and microscopic evidence of cure

SECONDARY OUTCOMES:
Physical examinations including examination of the muscles, joints, and bones; vital sign measurements, laboratory tests, and incidence of adverse events including any report of joint pain or joint disease

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Arguedas A, Dagan R, Pichichero M, Leibovitz E, Blumer J, McNeeley DF, Melkote R, Noel GJ. An open-label, double tympanocentesis study of levofloxacin therapy in children with, or at high risk for, recurrent or persistent acute otitis media. Pediatr Infect Dis J. 2006 Dec;25(12):1102-9. doi: 10.1097/01.inf.0000246828.13834.f9. PMID 17133154
- See also: A Study of Levofloxacin to Evaluate Bacteriologic Outcome in Children with Difficult To Treat Acute Otitis Media — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=477&filename=CR002389_CSR.pdf